CLINICAL TRIAL: NCT00517660
Title: Source Profiling of Biohazardous Aerosols in Hospitals
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Hong Kong University of Science and Technology (Other)
Other Study IDs: KC/KE-04-0071/ER-1; HARECCTR0500055
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Respiratory Tract Infections
Keywords: Healthy subjects; Lower Respiratory Tract Infections; Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
To characterise the physical parameters (number concentration, size distribution and their trajectories) of aerosols (droplets) generated in high risk procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years old) that can give valid consent
2. URTI: with symptoms such as coryza, sore throat, nasal discharge, cough and sputum +/- fever. Amongst these, cough should be a major complaint.
3. LRTI (CAP): acute lower respiratory illness of no other known cause which is usually associated with fever, symptoms and signs of the chest and abnormalities on the CXR. (BTS 1993).

Exclusion Criteria:

1. Pneumonia developed at or after 48 hours, or history of hospital admissions within 1 month of the present admission (to exclude hospital-acquired infections)
2. Patients who are unable to cooperate with the study protocols (such as mentally confused, dementia) or are physically unable to sit or stand independently to carry out the tests optimally.
3. Patients with TOCC associations with infections such Avian Flu or SARS (travel to endemic areas, at-risk occupations, close contacts with index cases, especially with compatible clinical features) or NPA revealed positivity of influenza A/B
4. Patients who are clinically or haemodynamically unstable, such as the need for inotropes, oxygen supplement of >2L/min, any types of shock, etc.
5. Underlying diseases that might affect the coughing effort (such as musculoskeletal diseases, or severe kyphoscoliosis)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 from each groups. Healthy subjects - recruited from voluntary basis. LRTI - recruited from patient wards with consent. URTI - recruited from out-patient clinic with consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-03; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Fang, Prof, Principal Investigator — Institute for the Environment, The Hong Kong University of Science and Technology
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, China